CLINICAL TRIAL: NCT03297567
Title: Control Group, Randomized, Blind Assessment of Physical Therapy Guidelines For Hospitalized Elderly
Brief Title: Physical Therapy Guidelines For Hospitalized Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Cidade de Sao Paulo (Other)
Responsible Party: Principal Investigator, Adriana Claudia Lunardi, Principal Investigator, Universidade Cidade de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 970669320241192
Record Dates: First submitted 2017-09-21; First posted 2017-09-29 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Physical Activity; Hospitalization; Aged; Exercise
Keywords: Elderly; Hospitalization; Immobilization; Exercise; Accelerometry
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: The patients will be randomized into two groups: intervention and control. The intervention group will receive verbal guidance and a booklet developed by the authors on the deleterious effects of hospitalization and the importance of staying active during hospital admission on the day they are included in the study. The control group will not receive any type of intervention, nor even verbal guidance.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigations of the level of physical activity, functional outcome, peripheral muscle strength and clinical complications will be performed by a blind investigator. Data analysis will be performed by a blind investigator in the control and intervention groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- verbal guidance and booklet (Experimental): verbal guidance and a booklet on the importance and benefits of movement during hospital stay, as well as what the patients should do to increase the level of physical activity.
  Interventions: Behavioral: verbal guidance and a booklet
- No Intervention (No Intervention): The control group will not receive any type of intervention

INTERVENTIONS:
Behavioral: verbal guidance and a booklet — Patients allocated to the intervention group will receive verbal instruction from the researchers on the importance and benefits of movement during hospital stay, as well as what they should do to increase the level of physical activity. These patients will receive the same guidelines through a playable, easy-to-understand and inexpensive booklet developed by the researchers themselves in PowerPoint 2016 (Microsoft) in order to remedy any doubt or forgetfulness during the hospitalization period
  Arms: verbal guidance and booklet

SUMMARY:
Introduction: The level of physical activity decreases progressively with age. Elderly subjects who are physically active have lower rates of morbidity and mortality when compared to those inactive. Hospitalization leads to long periods of bed rest and physical inactivity, with consequent muscle atrophy, generalized weakness, and decreased independence and functionality. Therefore, preventing inactivity, loss of muscle strength and the worsening of functional performance during hospitalization may be a way to avoid loss of independence. And while movement has been increasingly promoted as an important part of the recovery of hospitalized patients, many of them still spend much of the time bedridden while in hospital. Objectives: To evaluate the impact of a guiding program on the importance of remaining active during hospitalization in relation to the level of physical activity, functionality and muscular strength of elderly patients and to identify the main barriers that impede them to perform physical activities in the hospital environment. Methods: Randomized and controlled trial which will include elderly patients admitted to the Respiratory Diseases and Medical Clinic wards of the Institute of Medical Assistance to State Public Servants, in São Paulo. The intervention group will receive verbal guidelines and one booklet on the deleterious effects of hospitalization and the importance of staying active during hospitalization. All patients will be evaluated through accelerometry to identify the level of physical activity during hospitalization. Functionality will be evaluated through the DEMMI scale, muscular strength through handgrip and the main barriers to stay active during hospitalization by applying a questionnaire. The days of hospitalization and the clinical complications presented by the patients during the stay in the hospital will be noted. The difference of the outcomes of the level of physical activity and functionality before and after the intervention will be compared between the control and the intervention group through a t-test. The length of hospital stay will be analyzed by the Kaplan-Meier test and the incidence of complications by the chi-square test.

DETAILED DESCRIPTION:
Experimental Design: Patients located during the study period and who meet the eligibility criteria will be invited to participate and, after signing the informed consent form, will be evaluated for anthropometric and clinical characteristics. At this moment, patients will be randomized into two groups: intervention and control. The intervention group will receive verbal guidance and a booklet developed by the authors on the deleterious effects of hospitalization and the importance of staying active during hospital admission on the day they are included in the study. The control group will not receive any type of intervention, nor even verbal guidance. Patients from both groups will have an accelerometer placed on the wrist in the dominant limb, which should only be removed at hospital discharge. Besides the level of physical activity, patients will be evaluated for functionality, peripheral muscle strength, length of hospital stay, and incidence of complications during the hospitalization period. The researchers will contact the patients via telephone within 72 hours after hospital discharge in order to apply a questionnaire for identification of the main barriers to stay active during hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Admitted in the last 48 hours to the Respiratory Diseases and Medical Clinic wards
* Patients should not present restrictions to leave the bed
* Patients should not present need for professional help or accompanying person for locomotion
* Patients should not present local restriction for the placement of accelerometers (skin infections, amputation or fracture in the dominant limb)
* Patients should not present contact or respiratory isolation
* Patients should not present difficulty in understanding the guidelines or evaluations

Exclusion Criteria:

* Patients requiring hospital transfer
* Patients in need of surgical intervention
* Patients who not use the accelerometer during the proposed evaluation period

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2017-09-30 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Level of physical activity | All patients will be followed for the duration of hospital stay, an expected average of 7 days
  This variable will be evaluated by means of accelerometry using the an ActiGraph accelerometer (Actigraph Inc, USA) placed on the wrist of the patient's dominant limb in the first 48 h of admission. The calibration will be performed 24 hours a day, during the entire period of hospitalization, and will be removed only at the moment of hospital discharge. The equipment is waterproof, so there is no need to remove it for bath or personal hygiene, and its battery lasts up to 20 days of consecutive collection. The Actigraph GT3X records the number of steps, the time in different body positions, the intensity of movements and predicts the metabolic rate

SECONDARY OUTCOMES:
Functionality | All patients will be followed for the duration of hospital stay, an expected average of 7 days
  The evaluation of functionality will be done by applying the Morton Mobility Index (DEMMI). The DEMMI is a validated scale for elderly individuals during hospitalization and evaluates 15 activities divided into 5 groups: activities in bed, in the chair, static balance, ambulation and dynamic balance. The examiner's evaluation consists in punctuating the performance of the elderly in each of the motor conditions with scores varying from 0.1 to 2 points, resulting in a maximum score of 19 points. A conversion table allows the transformation of the raw score into a specific scale score, called DEMMI scores, ranging from 0 to 100 points, with higher scores indicating a higher level of mobility. The DEMMI scale consists of a paper sheet to be filled with a ballpoint pen, with printed articles on one side and the instruction protocol on the other, which makes it easy to use in clinical practice.
Peripheral Muscular Strength | All patients will be followed for the duration of hospital stay, an expected average of 7 days
  This will be evaluated after inclusion of the patient in the study and at the time of hospital discharge by a handgrip dynamometer (Smedley, Sahean, Belgium). The examiner will position the patient sitting and reclining comfortably in a chair with his feet flat on the floor. The dominant upper limb of the patient should maintain a 90-degree flexion without support and forearm in a neutral position. The unexamined upper limb will be resting, with the hand resting on the thigh. The patient will be asked to perform the manual grip movement. This movement will be repeated three times, with one-minute rest between attempts. The average of the three attempts will be adopted, which will be analyzed in its absolute value and in the reference value previously described for the Brazilian population.
Length of hospital stay | All patients will be followed for the duration of hospital stay, an expected average of 7 days
  It will be counted from admission to the ward until discharge
Incidence of complications | All patients will be followed for the duration of hospital stay, an expected average of 7 days
  These will be checked until the day of discharge through the records of a doctor who will be blind to the group to which the patient belongs. Clinical complications, specifically the appearance of a new health condition during hospitalization will be reported.
Barriers to stay active during hospitalization | 72 hours after hospital discharge
  These will be evaluated within 72 hours after hospital discharge. A questionnaire developed by the researchers themselves and evaluated by specialists (physical therapists who work in the hospital area with more than five years of experience) will be applied via telephone contact. The questionnaire is composed of 16 dichotomous questions with "yes" or "no" answers. The questions concern the presented symptoms and the patient, the knowledge about the importance of the physical activity and the hospital. After the creation of the questionnaire, this was subjected to an evaluation of pertinence and understanding of the questions by 30 physical therapists who work in the hospital area and have at least 5 years of experience. All suggested modifications were accepted and the questionnaire will be applied to the patients.
Number of Physiotherapy sessions | All patients will be followed for the duration of hospital stay, an expected average of 7 days
  The number of physiotherapy sessions received by the patient during the hospitalization period will be counted through the physiotherapeutic evolutions.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Lunardi, Study Director — Universidade Cidade de Sao Paulo
Locations (1):
- Instituto de Assistência Médica ao Servidor Público Estadual, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moreno NA, de Aquino BG, Garcia IF, Tavares LS, Costa LF, Giacomassi IWS, Lunardi AC. Physiotherapist advice to older inpatients about the importance of staying physically active during hospitalisation reduces sedentary time, increases daily steps and preserves mobility: a randomised trial. J Physiother. 2019 Oct;65(4):208-214. doi: 10.1016/j.jphys.2019.08.006. Epub 2019 Sep 11. PMID 31521553